CLINICAL TRIAL: NCT03747250
Title: Videolaryngoscopy Versus Direct Laryngoscopy for Elective Airway Management in Pediatric Anesthesia: Randomized Controlled Trial
Brief Title: Videolaryngoscopy vs. Direct Laryngoscopy for Elective Airway Management in Pediatric Anesthesia
Acronym: Videoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KDAR FN Brno 2018/12
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-02

CONDITIONS: Tracheal Intubation Morbidity
Keywords: Videolaryngoscopy; Laryngoscopy; Tracheal intubation; Success rate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: The allocation to the group will be randomized in located in closed envelope, that will be opened in the operating theater before anesthesia induction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscopy (Experimental): Pediatric patients undergoing elective surgery with planned tracheal intubation for airway management. The tracheal intubation will be performed with the use of videolaryngoscope
  Interventions: Device: Videolaryngoscopy
- Direct laryngoscopy (Active Comparator): Pediatric patients undergoing elective surgery with planned tracheal intubation for airway management. The tracheal intubation will be performed with the use of direct laryngoscopy
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: Videolaryngoscopy — In experimental group (interventional group), patients will be intubated with the videolaryngoscope
  Arms: Videolaryngoscopy
Device: Direct laryngoscopy — In control group (active comparator group), patients will be intubated with the direct laryngoscope
  Arms: Direct laryngoscopy

SUMMARY:
Videolaryngoscopy can lead to superior airway conditions and to the possible higher success compared to standard direct laryngoscopy. Patient will be randomized to the interventional group (videolaryngoscopy) and control group (direct laryngoscopy). The first attempt success rate, time to first end-tidal CO2 (ETCO2) wave, overall success rate, incidence of aspiration, bradycardia, desaturation a overall complications will be monitored.

DETAILED DESCRIPTION:
Videolaryngoscopy is specialized equipment for airway management, where a camera located at the tip of the laryngoscope blade can visualize also structures that can´t be seen on direct laryngoscopy, co the operator can obtain superior view of aditus laryngis during intubation. Currently videolaryngoscopy is not routinely used for intubation and it is reserved for patients with difficult airway. The aim of the trial is to compare the elective use of videolaryngoscopy versus direct laryngoscopy for elective airway management (tracheal intubation). Patients after informed consent approval will be randomized to the interventional group (videolaryngoscopy) and control group (laryngoscopy). The randomization will be managed by the Institute of Biostatistics and Analyses by the Faculty of medicine, Masaryk university. The primary aim will be the first intubation attempt success rate, the secondary aims will be time to successful intubation (time to first ETCO2 wave), overall success rate, number of intubation attempts, incidence of aspiration, desaturation and incidence of overall complications in all operators, in trainees, residents (5-10 years of practice), consultants (10-15 years of clinical practice) and consultants with over 15 years of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for elective surgery
* Planned tracheal intubation for airway management during surgery
* Signed informed consent

Exclusion Criteria:

* Emergency surgery
* Other airway management plan
* age outside the predefined limits
* Informed consent not signed

Ages: 29 Days to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 501 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
First intubation attempt success rate | Intraoperatively
  Success rate of the first intubation attempt

SECONDARY OUTCOMES:
Time for successful intubation | Intraoperatively
  Time need for intubation from decision to intubate to first end-tidal CO2 wave
Overall intubation success rate | Intraoperatively
  Success rate fot intubation
Laryngeal view | Intraoperatively
  Laryngeal view scored by Cormack-Lehane grading system
Complications | Intraoperatively
  Incidence of associated complications during anesthesia induction - desaturation, bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, assoc.Prof.MD.Ph.D, Study Chair — KDAR FN Brno
Locations (1):
- University Hospital Brno - FN Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klabusayova E, Klucka J, Kosinova M, Toukalkova M, Stoudek R, Kratochvil M, Marecek L, Svoboda M, Jabandziev P, Urik M, Stourac P. Videolaryngoscopy vs. Direct Laryngoscopy for Elective Airway Management in Paediatric Anaesthesia: A prospective randomised controlled trial. Eur J Anaesthesiol. 2021 Nov 1;38(11):1187-1193. doi: 10.1097/EJA.0000000000001595. PMID 34560686